CLINICAL TRIAL: NCT04192214
Title: A Two Arm Randomised, Open-label Study to Investigate the Persistence of Autoantibody Neutralisation, the Safety, and Pharmacokinetics of BC 007 in Patients With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF) and Autoantibodies Directed Against the beta1 Adrenergic Receptor
Brief Title: The Persistence of Autoantibody Neutralisation by BC 007 in Patients With Chronic HFrEF and Autoantibodies Against the Beta1-Adrenergic Receptor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Berlin Cures GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBC007C201
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cardiomyopathy, Dilated; Heart Failure; Autoantibodies
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BC 007 (Active Comparator): The treatment arm will comprise 20 randomly allocated β1-AAb positive dilative cardiomyopathy (DCM) patients. Participants will receive a continuous 75 minute infusion of 1350 mg BC 007 at day 1. The β1-AAb status will be monitored 10 days after treatment and every month. Treatment is repeated once up to month 11 if the participant's β1-AAbs were not neutralized after 1st dosing on day 1 or reoccur.
  Interventions: Drug: BC 007
- Control (No Intervention): The control arm will comprise 10 randomly allocated β1-AAb positive DCM patients. Participants will receive standard therapy but no intervention. The β1- AAb status will be monitored every month.

INTERVENTIONS:
Drug: BC 007 — 1350 mg of BC 007
  Arms: BC 007

SUMMARY:
Chronic heart failure (CHF) is one of the major causes of death in Western societies. Evidence has accumulated that functionally active autoantibodies directed against the beta1 adrenergic receptor (β1 AAb) are of pathophysiological relevance for the development and progression of cardiomyopathy and associated CHF. BC 007 is under development for targeted neutralisation of autoantibodies directed against G protein coupled receptors, including β1 AAb. This is an open label, three-centre, randomised phase 2a study in participants with chronic HFrEF. The study will evaluate whether BC 007 causes a persistent neutralisation of the β1 AAb demonstrated by a negative β1 AAb status up to 12 months. Participants will be randomised in a 2:1 ratio to the treatment arm (BC 007) or the control arm (untreated). Treatment is repeated once up to month 11 if the participant's β1 AAb were not neutralised after 1st dosing on day 1 or reoccur.

DETAILED DESCRIPTION:
Primary objective is:

- To compare the efficacy of an intravenous (i.v.) infusion of BC 007 with an untreated control arm in removal of β1 AAb at month 12 in participants with chronic heart failure with reduced ejection fraction (HFrEF)

Secondary objectives are:

* To evaluate the time to recurrence of β1 AAb after a single i.v. infusion of BC 007
* To evaluate the response rate and time to recurrence of β1 AAb after a repeated single i.v. infusion of BC 007 after the first recurrence of β1 AAb
* To evaluate the safety and tolerability of BC 007 after a single and a repeated single i.v. infusion
* To determine the pharmacokinetic (PK) plasma and urine profiles of BC 007
* To investigate the PK plasma profiles of BC 007 metabolites
* To investigate the β aminoisobutyric acid (β-AIBA) plasma and urine, and uric acid serum and urine concentration as a marker for BC 007 degradation
* To investigate the spontaneous conversion of β1 AAb status from positive to negative in untreated participants (control arm)

Exploratory objective is:

- To evaluate the change of the left ventricular ejection fraction (LVEF) after a single and a repeated single i.v. infusion

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant ≥18 years of age, at the time of signing the informed consent.
* Participant has CHF class II III, according to the NYHA classification.
* Participant has a chronic HFrEF with a left ventricular ejection fraction (LVEF) ≤40 % during screening (as assessed by in-hospital echocardiography).
* Participant screened positive for β1 AAb by a validated functional assay.

Exclusion Criteria:

* Participant has a sustained systolic blood pressure ≥160 mmHg prior to randomisation.
* Participant has a sustained bradycardia with resting heart rate <45 beats per minute (bpm) or tachycardia with resting heart rate >100 bpm prior to randomisation.
* Participant has an untreated primary valvular disease, considered clinically significant by the Investigator.
* Participant has any condition or therapy, which would make the participant unsuitable for the study, or life expectancy less than 12 months (e.g., active malignancy).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Proportion of β1 AAb negative participants at month 12 | 12 month

SECONDARY OUTCOMES:
Persistence of response defined as the time from initial β1 AAb neutralisation to β1 AAb recurrence. | 12 month
Response rate defined as the percentage of β1 AAb negative participants after a second treatment and persistence of response defined as the time from subsequent β1 AAb neutralisation to β1 AAb recurrence | 12 month
Comparative conversion rate of β1 AAb from positive to negative status measured by a cardiomyocyte beat rate assay in untreated participants (control arm) | 12 month
Number of Participants with abnormal laboratory values and/or adverse events that are related to treatment | 12 month
Area under the plasma concentration time curve (AUC) from time zero to the last quantifiable concentration (AUC0-t) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Area under the plasma concentration time curve (AUC) from time zero extrapolated to infinity (AUC0-inf) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Maximum observed plasma concentration (Cmax) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Apparent terminal half-life (t1/2) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Nominal time of Cmax (tmax) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Plasma clearance (CL) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Volume of distribution during terminal phase (Vz) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Terminal elimination rate constant (λz) derived from BC 007 and BC 007 metabolite (N-1, N-2 and N-3) plasma concentrations | 6 hour post start of infusion
Cumulative amount of unchanged drug excreted into urine (Ae) | 6 hour post start of infusion
Fraction of intravenous administered drug that is excreted unchanged in urine (fe) | 6 hour post start of infusion
Renal clearance (CLR) of BC 007 | 6 hour post start of infusion
Area under the plasma concentration time curve (AUC) from time zero to the last quantifiable concentration (AUC0-t) derived from β-aminoisobutyric acid and uric acid plasma concentrations | 6 hour post start of infusion
Area under the plasma concentration time curve (AUC) from time zero to the concentration after 4 hours (AUC0-4h) derived from β-aminoisobutyric acid and uric acid plasma concentrations | 4 hour post start of infusion
Area under the plasma concentration time curve (AUC) from time zero to the concentration after 6 hours (AUC0-6h) derived from β-aminoisobutyric acid and uric acid plasma concentrations | 6 hour post start of infusion
Area under the plasma concentration time curve (AUC) from time zero extrapolated to infinity (AUC0-inf) derived from β-aminoisobutyric acid and uric acid plasma concentrations | 6 hour post start of infusion
Maximum observed plasma concentration (Cmax) derived from β-aminoisobutyric acid and uric acid plasma concentrations | 6 hour post start of infusion
Nominal time of Cmax (tmax) derived from β-aminoisobutyric acid and uric acid plasma concentrations | 6 hour post start of infusion
Cumulative amount of β-aminoisobutyric acid and uric acid excreted into urine (Ae) | 6 hour post start of infusion
Renal clearance (CLR) of β-aminoisobutyric acid and uric acid | 6 hour post start of infusion

OTHER OUTCOMES:
Echocardiographic parameter LVEF compared to untreated participants (control arm) from baseline to month 12 | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Müller, Dr., Study Director — Berlin Cures GmbH
Locations (3):
- Serbia (3):
  - Bežanijska Kosa Clinical and Hospital Centre, Belgrade
  - Institut za kardiovaskularne bolesti Dedinje, Belgrade
  - Zvezdara Clinical and Hospital Centre, Belgrade

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haberland A, Holtzhauer M, Schlichtiger A, Bartel S, Schimke I, Muller J, Dandel M, Luppa PB, Wallukat G. Aptamer BC 007 - A broad spectrum neutralizer of pathogenic autoantibodies against G-protein-coupled receptors. Eur J Pharmacol. 2016 Oct 15;789:37-45. doi: 10.1016/j.ejphar.2016.06.061. Epub 2016 Jul 1. PMID 27375076
- [Background] Wenzel K, Schulze-Rothe S, Haberland A, Muller J, Wallukat G, Davideit H. Performance and in-house validation of a bioassay for the determination of beta1-autoantibodies found in patients with cardiomyopathy. Heliyon. 2017 Jul 31;3(7):e00362. doi: 10.1016/j.heliyon.2017.e00362. eCollection 2017 Jul. PMID 28795160
- [Background] Wallukat G, Muller J, Haberland A, Berg S, Schulz A, Freyse EJ, Vetter R, Salzsieder E, Kreutz R, Schimke I. Aptamer BC007 for neutralization of pathogenic autoantibodies directed against G-protein coupled receptors: A vision of future treatment of patients with cardiomyopathies and positivity for those autoantibodies. Atherosclerosis. 2016 Jan;244:44-7. doi: 10.1016/j.atherosclerosis.2015.11.001. Epub 2015 Nov 10. PMID 26584137